CLINICAL TRIAL: NCT06803914
Title: Analysis of Biomechanical Parameters and Return to Sport After Total Hip Replacement
Status: Recruiting | Type: Observational
Sponsor: Clinique du Sport, Bordeaux Mérignac (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-31-SBM
Record Dates: First submitted 2025-01-13; First posted 2025-01-31 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Hip Arthroplasty, Total

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Biomechanical analysis
  Interventions: Procedure: Biomechanical analysis

INTERVENTIONS:
Procedure: Biomechanical analysis — Biomechanical assessment is performed using a set of sensors (Qualisys Sports Marker Set - functional assessment, already in use at the Clinique du Sport) as well as 3D optoelectronic cameras and force and pressure platforms. These sensors are placed at various points on both lower limbs (hip, knee, ankle) and provide data in different planes (sagittal, frontal, transverse), as well as a comparison of both sides.

SUMMARY:
This prospective study aims to evaluate the dynamic biomechanical parameters of gait in active patients who have undergone total hip replacement (THR), focusing on movements critical for return to sport.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for total hip replacement surgery
* Active patient with low to high level of physical activity prior to surgery
* Informed consent
* Complete medical file

Exclusion Criteria:

* Contralateral hip surgery
* Neurological disorder affecting movement (e.g. Parkinson's disease, stroke)
* Spinal pathology affecting movement or posture
* Dementia or inability to complete questionnaires and assessments
* Pregnant or breast-feeding patient
* Patient under protective supervision
* Patient not covered by a social security scheme

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Active patients (low to high level of physical activity priori to surgery) with hip osteoarthritis necessiting total hip replacement
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Angular measurements by biomechanical sensors | 6 months after surgery
  Angle measurements at hip, pelvis, knee and ankle in the three planes of space (sagittal, frontal and transverse), measured by biomechanical sensors.
Vertical forces measured by biomechanical sensors | 6 months after surgery
  Vertical forces, push and landing, will be evaluated for each phase of the movements. Biomechanical specific sensors will be used to measure these data

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique du Sport, Mérignac, France

IPD SHARING:
Plan to Share IPD: No